CLINICAL TRIAL: NCT01958047
Title: A Phase 1 Open-label Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a Single Dose of ASP3652 in Caucasian, Japanese, Black/African and Chinese Healthy Male and Female Subjects
Brief Title: A Study to Assess the Effect of Race on How a Single Dose of ASP3652 is Taken up, Metabolized and Distributed Through the Bodies of Young, Healthy Male and Female Subjects, and Its Safety and Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3652-CL-0054; 2012-001476-11 (EudraCT Number)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Pharmacokinetics; Pharmacodynamics; Healthy Subjects; Effect of Race
Keywords: Phase I; ASP3652; Single dose; Dietary intake
MeSH Terms: interventions — ASP3652

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP3652 (Experimental): One single dose
  Interventions: Drug: ASP3652

INTERVENTIONS:
Drug: ASP3652 — Oral

SUMMARY:
This study investigates how ASP3652 is taken up, broken down, and distributed through the body and excreted in individuals of different races. The study also investigates levels of biochemical markers in the bloodstream, and determines how safe the study drug is and how well it is tolerated after dosing. A further aim is to look at how the processes of metabolism, distribution and excretion of the study drug are possibly altered by the daily diet of the volunteers taking part.

DETAILED DESCRIPTION:
This is an open label study to assess the pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability of a single dose of ASP3652 in healthy male and female subjects from Caucasian, Japanese, Black/African and Chinese origin.

A total of 64 healthy male and female subjects are included in this study (16 subjects per race group). Each race group comprises 8 female subjects and 8 male subjects.

Screening assessments are performed from Day -22 to Day -2, and subjects are admitted to the clinic on Day -1, where they remain until Day 4. On Day 1, the subjects receive a single oral dose of ASP3652, and are discharged on Day 4 when all assessments have been performed and if there are no medical reasons to stay longer. An end of study visit (ESV) is performed 7-14 days after discharge.

For each race group, plasma samples for PK and PD analysis are collected. Vital signs, safety electrocardiogram (ECG) measurements, safety laboratory assessments, physical examination, adverse events (AEs) and concomitant medications are monitored throughout study.

In order to identify potential relationships between dietary intake and the PK of a single dose of ASP3652, all subjects record their diet for 3 days during the screening period in order to assess daily dietary intake (including total daily caloric intake; daily cholesterol intake; and total fat, saturated fat, carbohydrate and protein as a percentage of total calories).

ELIGIBILITY:
Inclusion Criteria:

* The subject is a healthy male or female subject from Caucasian, Japanese, Black/African or Chinese origin. Both parents and all 4 grandparents should be of the same race.
* Subjects of Japanese or Chinese origin should be born in their respective countries and should not have lived outside of their countries for more than 5 years and 10 years, respectively.
* The subject has a Body Mass Index (BMI) in the range 18.5 - 30.0 kg/m2, inclusive (subject from Caucasian or Black/African origin) or in the range 17.5 - 29.0 kg/m2, inclusive (subject from Japanese or Chinese origin). The subject weighs at least 50 kg (subject from Caucasian or Black/African origin) or at least 45 kg (subject from Japanese or Chinese origin).

Exclusion Criteria:

* Female subject who is pregnant, has been pregnant within 6 months before screening, or breast feeding within 3 months before screening.
* Known or suspected hypersensitivity to ASP3652 or any components of the formulation used.
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to admission to the Clinical Unit.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP3652 in plasma measured by Cmax | Day 1 to Day 4 (16 blood samples taken)
  maximum observed plasma concentration (Cmax)
Pharmacokinetics of ASP3652 in plasma measured by AUClast | Day 1 to Day 4 (16 blood samples taken)
  area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast)
Pharmacokinetics of ASP3652 in plasma measured by AUCinf | Day 1 to Day 4 (16 blood samples taken)
  area under the plasma concentration-time curve from time zero extrapolated to the infinite time (AUCinf)
Pharmacokinetics of ASP3652 in plasma measured by tmax | Day 1 to Day 4 (16 blood samples taken)
  time to attain Cmax (tmax)
Pharmacokinetics of ASP3652 in plasma measured by tlag | Day 1 to Day 4 (16 blood samples taken)
  PK lag time (tlag)
Pharmacokinetics of ASP3652 in plasma measured by t1/2 | Day 1 to Day 4 (16 blood samples taken)
  apparent terminal elimination half-life (t1/2)
Pharmacokinetics of ASP3652 in plasma measured by Vz/F | Day 1 to Day 4 (16 blood samples taken)
  apparent volume of terminal phase distribution at steady state (Vz/F)
Pharmacokinetics of ASP3652 in plasma measured by CL/F | Day 1 to Day 4 (16 blood samples taken)
  apparent clearance after oral administration at steady state (CL/F)
Pharmacokinetics of ASP3652 in plasma measured by Vz/F/kg | Day 1 to Day 4 (16 blood samples taken)
  body weight-adjusted apparent volume of terminal phase distribution at steady state (Vz/F/kg)
Pharmacokinetics of ASP3652 in plasma measured by CL/F/kg | Day 1 to Day 4 (16 blood samples taken)
  body weight-adjusted apparent clearance after oral administration at steady state (CL/F/kg)
Pharmacokinetics of ASP3652 metabolites in plasma measured by Cmax | Day 1 to Day 4 (16 blood samples taken)
Pharmacokinetics of ASP3652 metabolites in plasma measured by AUClast | Day 1 to Day 4 (16 blood samples taken)
Pharmacokinetics of ASP3652 metabolites in plasma measured by AUCinf | Day 1 to Day 4 (16 blood samples taken)
Pharmacokinetics of ASP3652 metabolites in plasma measured by tmax | Day 1 to Day 4 (16 blood samples taken)
Pharmacokinetics of ASP3652 metabolites in plasma measured by tlag | Day 1 to Day 4 (16 blood samples taken)
  tlag
Pharmacokinetics of ASP3652 metabolites in plasma measured by t1/2 | Day 1 to Day 4 (16 blood samples taken)

SECONDARY OUTCOMES:
Plasma levels of arachidonoyl-ethanolamide (AEA, or anandamide), oleoyl-ethanolamide (OEA) and palmitoyl-ethanolamide (PEA) after a single dose of ASP3652 | Day 1 to Day 4 (12 blood samples taken)
  maximum response (Rmax), time of the maximum response (tmax R), area under the response curve (AUR)
Safety and tolerability of a single dose of ASP3652 | Screening to ESV (at least 39 safety assessments)
  vital signs, safety electrocardiogram measurements, safety laboratory assessments, physical examination and adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Clincial Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, United Kingdom